CLINICAL TRIAL: NCT04518280
Title: A Prospective Phase II Trial of Short-course Radiotherapy Based Total Neoadjuvant Therapy Combined With PD-1 Inhibitor for Locally Advanced Rectal Cancer (TORCH）
Brief Title: Short-course Radiotherapy Based TNT Combined With PD-1 Inhibitor for Locally Advanced Rectal Cancer
Acronym: TORCH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhen Zhang, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FDRT-2020-236-2156
Record Dates: First submitted 2020-08-15; First posted 2020-08-19 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Locally Advanced Rectal Cancer
MeSH Terms: interventions — spartalizumab; toripalimab; Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): The patients will receive short-course radiotherapy (25Gy/5Fx), followed by 6 cycles of CAPOX and PD-1 antibody. TME surgery is scheduled after TNT while a W&W option can be applied to patients achieving cCR.
  Interventions: Drug: PD-1 antibody; Drug: Capecitabine; Drug: Oxaliplatin; Radiation: Short-course radiotherapy
- Group B (Experimental): The patients will firstly receive 2 cycles of CAPOX and PD-1 antibody, then receive short-course radiotherapy (25Gy/5Fx), followed by 4 cycles of CAPOX and PD-1 antibody. TME surgery is scheduled after TNT while a W&W option can be applied to patients achieving cCR.
  Interventions: Drug: PD-1 antibody; Drug: Capecitabine; Drug: Oxaliplatin; Radiation: Short-course radiotherapy

INTERVENTIONS:
Drug: PD-1 antibody — PD-1 antibody (Toripalimab): 240mg d1 q3w
  Other Names: Toripalimab
Drug: Capecitabine — Capecitabine: 1000mg/m2 bid d1-14 q3w
  Other Names: Xeloda
Drug: Oxaliplatin — Oxaliplatin: 130mg/m2 d1 q3w
Radiation: Short-course radiotherapy — Shor-course radiotherapy: 25Gy/5Fx

SUMMARY:
TORCH is a prospective, multicentre, randomized phase II trial. 130 LARC (T3-4/N+M0, distance from anal verge ≤12cm) patients will be treated with total neoadjuvant therapy (TNT) and assigned to Group A and Group B. Group A receives SCRT (25Gy/5Fx) followed by 6 cycles of Toripalimab combined with CAPOX (ToriCAPOX). Group B receives 2 cycles of ToriCAPOX followed by SCRT and 4 cycles of ToriCAPOX. TME surgery is scheduled after TNT while a watch and wait (W&W) option can be applied to patients achieving clinical complete response (cCR). The primary endpoint is complete response (CR, pathological complete response [pCR] plus cCR) rate. The secondary endpoints include the grade 3-4 acute adverse effects (AE) rate, 3-year DFS rate, etc.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological confrmed adenocarcinoma
2. Clinical stage T3-4 and/or N+
3. The distance from anal verge ≤12 cm
4. Without distance metastases
5. Age 18-70 years old, female and male
6. KPS > =70
7. Baseline blood and biochemical indicators meet the following criteria: neutrophils≥1.5×10^9/L, Hb≥90 g/L, PLT≥100×10^9/L, ALT/AST≤2.5 ULN, Cr≤1 ULN
8. With good compliance and signed the consent form

Exclusion Criteria:

1. Pregnancy or breast-feeding women
2. Known history of other malignancies within 5 years
3. Known history of previous anti-tumor treatment, including radiotherapy, chemotherapy, immune checkpoint inhibitors, T cell-related therapy, etc
4. Known history of severe neurological or mental illness (such as schizophrenia, dementia or epilepsy)
5. Current severe cardiac disease (cardiac dysfunction and arrhythmia), renal dysfunction and liver dysfunction
6. Acute cardiac infarction or cerebral ischemic stroke occurred within 6 months before recruitment
7. Uncontrolled infection which needs systemic therapy
8. Active autoimmune disease or immunodefciencies, known history of organ transplantation or systematic use of immunosuppressive agents
9. Known history of human immunodefciency virus (HIV) infection (i.e., HIV 1 to 2 antibody positive), active syphilis infection, active pulmonary tuberculosis infection
10. Active Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening (i.e., HBsAg positive or HBV DNA positive, HCV RNA positive if anti-HCV antibody testing positive)
11. Allergic to any component of the therapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Complete response (CR) rate | The status of cCR will be evaluated after the completion of neoadjuvant therapy. The pCR rate will be evaluated after surgery. The cCR patients who adopted W&W strategy will be included into the CR rate caluculation.
  Rate of complete response (CR), including the rate of pathologic complete response (pCR) after surgery and the rate of cCR with W&W strategy.

SECONDARY OUTCOMES:
Grade 3-4 adverse effects rate | From date of randomization until the date of death from any cause, assessed up to 5 years
  Rate of chemotherapy, radiotherapy and immunotherapy related adverse events
3 year disease free survival rate | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months.
  Rate of 3 year disease free survival
3 year local recurrence free survival rate | From date of randomization until the date of first documented pelvic failure, assessed up to 36 months.
  Rate of 3 year local recurrence free survival
3 year overall survival rate | From date of randomization until the date of death from any cause, assessed up to 36 months.
  Rate of 3 year overall survival
Rate of Surgical complications | The surgery was scheduled 2-4 weeks after the end of neoadjuvant therapy. And the surgical complications were assessed up to 5 years from the surgery.
  Rate of surgical complications, such as intraoperative hemorrhage, anastomotic leakage, intestinal obstruction, etc.
Scores of Quality of Life | From date of randomization until the date of death from any cause, assessed up to 10 years
  Quality of life will be evaluated using EORTC QLQ-C30, EORTC QLQ-CR29, LARS score and Wexner score.

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Zhang, M.D, PH.D, Principal Investigator — Fudan University
Locations (3):
- China (3):
  - Shanghai Changhai Hospital, Shanghai, Shanghai Municipality
  - Zhen Zhang, Shanghai, Shanghai Municipality
  - Shanghai East Hospital, Shanghai

REFERENCES:
- [Derived] Xia F, Wang Y, Wang H, Shen L, Xiang Z, Zhao Y, Zhang H, Wan J, Zhang H, Wang Y, Wu R, Wang J, Yang W, Zhou M, Zhou S, Chen Y, Zhang Z, Wu X, Xuan Y, Wang R, Sun Y, Tong T, Zhang X, Wang L, Huang D, Sheng W, Yan H, Yang X, Shen Y, Xu Y, Zhao R, Mo M, Cai G, Cai S, Xu Y, Zhang Z. Randomized Phase II Trial of Immunotherapy-Based Total Neoadjuvant Therapy for Proficient Mismatch Repair or Microsatellite Stable Locally Advanced Rectal Cancer (TORCH). J Clin Oncol. 2024 Oct;42(28):3308-3318. doi: 10.1200/JCO.23.02261. Epub 2024 Jul 1. PMID 38950321
- [Derived] Wang Y, Shen L, Wan J, Zhang H, Wu R, Wang J, Wang Y, Xu Y, Cai S, Zhang Z, Xia F. Short-course radiotherapy combined with CAPOX and Toripalimab for the total neoadjuvant therapy of locally advanced rectal cancer: a randomized, prospective, multicentre, double-arm, phase II trial (TORCH). BMC Cancer. 2022 Mar 15;22(1):274. doi: 10.1186/s12885-022-09348-z. PMID 35291966
- See also: TORCH JCO 2024 — https://pubmed.ncbi.nlm.nih.gov/38950321/